CLINICAL TRIAL: NCT05441085
Title: Programmed Intermittent Epidural Bolus Interval 90 Min of 10ml,0.0625% Bupivacaine Plus 2μg/mL Fentanyl in Nulliparous Versus Multiparous Parturient
Brief Title: Programed Intermittent Epidural Bolus Interval 90 (EI90) of 10 ml, 0.0625% Bupivacaine Plus 2 μg/mL Fentanyl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, rabab Mohammad habeeb, Principal investigator, Menoufia University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANET2022
Record Dates: First submitted 2022-06-22; First posted 2022-07-01 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Labour Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nulliparous (Active Comparator): Patients of ASA physical status 2-3 with a singleton pregnancy; gestational age > 37 weeks; regular uterine contractions occurring at least every 5 min; cervical dilation 2-5 cm; and pain > 5
  Interventions: Device: programed intermittent epidural bolus interval 90 (EI90)
- Multiparous (Active Comparator): Patients of ASA physical status 2-3 with a singleton pregnancy; gestational age > 37 weeks; regular uterine contractions occurring at least every 5 min; cervical dilation 2-5 cm; and pain > 5
  Interventions: Device: programed intermittent epidural bolus interval 90 (EI90)

INTERVENTIONS:
Device: programed intermittent epidural bolus interval 90 (EI90) — programed intermittent epidural bolus interval 90 (EI90) of 10 ml, 0.0625% bupivacaine plus 2 μg/mL fentanyl

SUMMARY:
Multiple studies showed the numerous advantages of implementing programmed epidural bolus (PIEB) technique, where a fixed volume of local anesthetic is automatically administrated at a set time interval compared to the continuous epidural infusion technique (CEI). The advantages were improved maternal satisfaction, decreased local anesthetic consumption, and decreased second stage of labor.The theory behind PIEB is that to attain a more uniform spread of local anesthetic in the epidural space a higher volume of injectate and a higher pressure is needed.Different approaches using different timings and volumes for PIEB have been proposed to achieve the optimal regimen. Many studies showed evidence that 10 mL boluses of bupivacaine 0.0625% with fentanyl 2 μg/mL delivered every 40 min, named effective programed intermittent epidural bolus interval 90 (EI90), produced effective analgesia without breakthrough pain in 90% of nulliparous women during the first stage of labor.

ELIGIBILITY:
Inclusion Criteria:

* Patients of ASA physical status 2-3 with a singleton pregnancy
* gestational age > 37 weeks
* regular uterine contractions occurring at least every 5 min;
* cervical dilation 2-5 cm
* pain > 5 (Visual analogue score (VAS) 0-10) at the time of request for epidural analgesia .

Exclusion Criteria:

* Refusal to concent
* Contraindication to epidural analgesia as allergy or hypersensitivity to bupivacaine or fentanyl
* Patients who had opioids or sedatives within 4 h preceding epidural insertion.
* Unintentional dural puncture.
* Patient who deliver within 1 h after initiation of epidural clinician bolus.
* The inability to achieve as VAS score ≤2 after the initial loading dose will be considered as a failure and will be excluded from the study.

Max Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Nulliparous and multiparous women
Enrollment: 30 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
adequate labour analgesia | six hours
  Time of first call for bolus dose of epidural After loading dose

SECONDARY OUTCOMES:
Upper sensory block | 24hours
  Secsensory block level to ice
Visual Analogue Scale to pain | 24 hours
  As zero is no pain and 10 is the maximum pain that can be felt
Motor block | 24 hours
  Motor block measured by bromage scale
Total anaesthetic volume | 24 hours
  Total volume of local anesthetic used
Side effects | 24 hours
  Presence of side effects as neusea, vomiting,peruritis

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Medicine Menoufia University, Cairo, Governorate
  - Rabab Habeeb, Cairo, Governorate

IPD SHARING:
Plan to Share IPD: No